CLINICAL TRIAL: NCT03318809
Title: A Phase 1, Open-label, Single-dose Study to Evaluate the Safety, Tolerability and Pharmacokinetics of AMG 986 Administered Orally to Healthy Volunteers and Subjects With Severely Impaired Renal Function
Brief Title: Study to Evaluate the Safety, Tolerability and Pharmacokinetics of AMG 986 Administered Orally to Healthy Volunteers and Participants With Severely Impaired Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20150186
Record Dates: First submitted 2017-10-06; First posted 2017-10-24 (Actual); Results first posted 2021-01-27 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-06

CONDITIONS: Heart Failure
Keywords: Cardiovascular Diseases; Renal Impairment; Heart Diseases
MeSH Terms: conditions — Heart Failure; Cardiovascular Diseases; Renal Insufficiency; Heart Diseases

STUDY DESIGN:
Intervention Model Description: This is a multisite (approximately 3 sites), open-label, non-randomized, single-dose study in participants with severely impaired kidney function and healthy participants. About 12 participants will be assigned to two groups: Group 1: 6 with severely impaired kidney function , and Group 2: 6 with normal kidney function.
Masking Description: The patient, investigator, investigative staff, medical monitor and care provider will not be masked for the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1: Severely Renal Impaired Participants (Experimental): Participants with severely impaired renal function (estimated glomerular filtration rate [eGFR] 15 to 29 mL/min/1.73 m^2) receive a single oral dose of 200 mg AMG 986.
  Interventions: Drug: AMG 986
- Group 2: Healthy Participants (Active Comparator): Participants with normal renal function (eGFR >= 90 mL/min/1.73 m^2 or above) receive a single oral dose of 200 mg AMG 986.
  Interventions: Drug: AMG 986

INTERVENTIONS:
Drug: AMG 986 — tablets for oral administration

SUMMARY:
A study to assess the safety, tolerability, and pharmacokinetics of AMG 986 given orally as a single dose to healthy participants and participants with severely impaired kidney function.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, who are > or = 18 and < or = 65 years of age at the time of screening
* Subject has provided informed consent prior to initiation of any study-specific activities/procedures
* Women must be of non-reproductive potential (ie, postmenopausal, history of hysterectomy, or history of bilateral oophorectomy)
* Men must agree to practice an acceptable method of effective birth control while on study through 11 weeks after receiving the dose of study drug.
* Men must be willing to abstain from sperm donation while on study through 11 weeks after receiving the dose of study drug
* Body Mass Index > or = 18 and < or = 38 kg/m^2 at screening
* Physical examination and 12-lead electrocardiograms (ECGs) are clinically acceptable to the investigator
* Non-hypertensive subjects or subjects with treated, stable hypertension as defined by blood pressure not exceeding 170/100 mm Hg as an average during screening and day -1; for subjects with renal impairment, no change in dosage and medication for > or = 4 weeks prior to screening, and expected to remain on this dose and medication for the entire duration of the study
* Willing to maintain current general diet and physical activity regimen
* Renal function in 1 of the following 2 categories at the time of screening: Group 1 - Severe Renal Impairment (eGFR 15 to 29 mg/min/1.73 m^2) and not anticipated to require hemodialysis or renal transplantation, and anticipated to have renal function appropriate to severe renal impairment for the duration of the study OR Group 2 - Normal renal function (eGFR > or = 90 mg/min/1.73 m^2)

Exclusion Criteria:

* Subjects whose second modification of diet in renal disease (MDRD) eGFR result on day -1 is not within 15% of the first eGFR result performed during the screening period. Healthy volunteers who have normal renal function, but show a difference greater than 15% in eGFR based on MDRD during the screening period, will be included in the trial at the discretion of the investigator and the sponsor after a 24-hour creatinine clearance has been performed that meets eligibility criteria.
* Subjects who are the recipient of a renal transplant and/or are on immunosupressants.
* Subjects with a history of hospitalization for heart disease or angina within 4 months of screening.
* Current or prior malignancy within 5 years of enrollment with the exception of non-melanoma skin cancers, cervical or breast ductal carcinoma in situ, and adenocarcinoma of the prostate Stage I or IIa (defined as T1, T2a or T2b, N0-, M0 with documented serum prostate-specific antigen (PSA) < 20 ng/mL and Gleason score ≤ 7) per the American Joint Committee on Cancer (AJCC) primary tumor, regional lymph nodes, and distant metastasis system.
* Positive for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg) or hepatitis C virus antibodies (HepCAb) at screening
* History or evidence of any other clinically significant disorder, condition or disease with the exception of those outlined above that, in the opinion of the investigator or Amgen physician, if consulted, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion.
* Subject previously has entered this study or has been previously exposed to AMG 986.
* Heart rate ≥ 100 beats per minute after 5 minutes of rest or an untreated symptomatic bradyarrhythmia within 1 month prior to enrollment.
* Known history of drug or alcohol abuse within last 12 months.
* Currently receiving treatment in another investigational device or drug study or less than 30 days or 5 half-lives (whichever is longer) since ending treatment on another investigational device or drug study(s) prior to receiving the dose of investigational product (AMG 986).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2018-03-12 (Actual); Study Completion 2018-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (4):
- United States (4):
  - Research Site, Tustin, California
  - Research Site, Orlando, Florida
  - Research Site, Minneapolis, Minnesota
  - Research Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication (or other new use) have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors, and if not approved, may be further arbitrated by a Data Sharing Independent Review Panel. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the link below.
URL: https://www.amgen.com/datasharing

REFERENCES:
- [Background] Trivedi A, Mather O, Vega S, Simiens MA, Hellawell J, Lee E. Effect of Severe Renal Impairment on the Safety, Tolerability, and Pharmacokinetics of AMG 986. Drugs R D. 2022 Mar;22(1):89-94. doi: 10.1007/s40268-021-00380-1. Epub 2022 Jan 29. PMID 35092583
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted in 4 centers in the United States.
Groups:
- Group 1: Severely Renal Impaired Participants: Participants with severely impaired renal function (estimated glomerular filtration rate [eGFR] 15 to 29 mL/min/1.73 m^2) received a single oral dose of 200 mg AMG 986.
- Group 2: Healthy Participants: Participants with normal renal function (eGFR >= 90 mL/min/1.73 m^2 or above) received a single oral dose of 200 mg AMG 986.
Period: Overall Study
Arm/Group | Group 1: Severely Renal Impaired Participants | Group 2: Healthy Participants
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all study participants who received at least 1 dose of AMG 986.
Groups:
- Group 1: Severely Renal Impaired Participants: Participants with severely impaired renal function (eGFR 15 to 29 mL/min/1.73 m^2) received a single oral dose of 200 mg AMG 986.
- Total: Total of all reporting groups
Arm/Group | Group 1: Severely Renal Impaired Participants | Group 2: Healthy Participants | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.7 (8.1) | 57.8 (3.3) | 57.3 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 6 | 5 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 1 | 1 | 2
  Black (or African American) | 3 | 3 | 6
  White | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: AMG 986 Pharmacokinetic (PK) Parameter: Area Under the Plasma Concentration Time Curve From Time 0 to the Time of the Last Quantifiable Sample (AUClast)
Time Frame: Predose, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120 hours post-dose
Population: The PK analysis set included all participants for whom at least 1 PK parameter or endpoint could be reliably estimated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Group 1: Severely Renal Impaired Participants | Group 2: Healthy Participants
Number analyzed (Participants) | 6 | 6
hr*ng/mL | 80,000 (33.6) | 64,500 (70.0)
Statistical Analysis 1: Comparison: Group 1: Severely Renal Impaired Participants vs Group 2: Healthy Participants; Test type: Other — Analysis of Variance; Ratio (Group 1/Group 2) = 1.24, 90% CI 2-sided [0.73 to 2.10] — The ratio and confidence interval (CI) are based on natural log scale data converted back to the original scale

2. Primary Outcome: AMG 986 PK Parameter: Maximum Observed Plasma Concentration After Dosing (Cmax)
Time Frame: 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120 hours post-dose
Population: The PK analysis set included all participants for whom at least 1 PK parameter or endpoint could be reliably estimated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Group 1: Severely Renal Impaired Participants | Group 2: Healthy Participants
Number analyzed (Participants) | 6 | 6
ng/mL | 10,600 (45.3) | 7520 (50.5)
Statistical Analysis 1: Comparison: Group 1: Severely Renal Impaired Participants vs Group 2: Healthy Participants; Test type: Other — Analysis of Variance; Ratio (Group 1/Group 2) = 1.41, 90% CI 2-sided [0.88 to 2.27] — The ratio and CI are based on natural log scale data converted back to the original scale

3. Primary Outcome: AMG 986 PK Parameter: Terminal Phase Half-Life (t1/2,z)
Time Frame: Predose, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120 hours post-dose
Population: The PK analysis set included all participants for whom at least 1 PK parameter or endpoint could be reliably estimated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Group 1: Severely Renal Impaired Participants | Group 2: Healthy Participants
Number analyzed (Participants) | 6 | 6
hours | 18.4 (21.1) | 21.1 (44.6)

4. Primary Outcome: AMG 986 PK Parameter: Time of Maximum Plasma Concentration (Tmax)
Time Frame: Predose, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120 hours post-dose
Population: The PK analysis set included all participants for whom at least 1 PK parameter or endpoint could be reliably estimated.
Measure: Median (Full Range); unit: hours
Arm/Group | Group 1: Severely Renal Impaired Participants | Group 2: Healthy Participants
Number analyzed (Participants) | 6 | 6
hours | 1.1 [1.0 to 2.1] | 1.5 [1.1 to 4.1]

5. Primary Outcome: AMG 986 PK Parameter: Area Under the Plasma Concentration Time Curve From Time 0 to Infinity (AUCinf)
Time Frame: Predose, 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120 hours post-dose
Population: The PK analysis set included all participants for whom at least 1 PK parameter or endpoint could be reliably estimated.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Group 1: Severely Renal Impaired Participants | Group 2: Healthy Participants
Number analyzed (Participants) | 6 | 6
ng*hr/mL | 80,800 (33.6) | 65,800 (68.8)
Statistical Analysis 1: Comparison: Group 1: Severely Renal Impaired Participants vs Group 2: Healthy Participants; Test type: Other — Analysis of Variance; Ratio (Group 1/Group 2) = 1.24, 90% CI 2-sided [0.73 to 2.10] — The ratio and CI are based on natural log scale data converted back to the original scale

6. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event is defined as any untoward medical occurrence in a clinical trial subject. A serious adverse event is defined as an adverse event that meets at least 1 of the following serious criteria:
  * fatal
  * life threatening (places the subject at immediate risk of death)
  * requires in patient hospitalization or prolongation of existing hospitalization
  * results in persistent or significant disability/incapacity
  * congenital anomaly/birth defect
  * other medically important serious event
Time Frame: From first dose of study drug up to Day 30
Population: The safety analysis set included all study participants who received at least 1 dose of AMG 986.
Measure: Number; unit: participants
Arm/Group | Group 1: Severely Renal Impaired Participants | Group 2: Healthy Participants
Number analyzed (Participants) | 6 | 6
participants
  TEAEs | 2 | 1
  Serious TEAEs | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to Day 30
Arm/Group | Group 1: Severely Renal Impaired Participants | Group 2: Healthy Participants
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 2/6 | 1/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: Severely Renal Impaired Participants (N=6) | Group 2: Healthy Participants (N=6)
Nausea (Gastrointestinal disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2017-09-28): https://cdn.clinicaltrials.gov/large-docs/09/NCT03318809/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-12): https://cdn.clinicaltrials.gov/large-docs/09/NCT03318809/SAP_001.pdf